CLINICAL TRIAL: NCT02214069
Title: Assessing the Accuracy of an Atrial Fibrillation Detection Algorithm Using Novel Smart Phone Technology in Detecting the Presence of Atrial Fibrillation. iRead Study
Brief Title: Using Smart Phone Technology in Detecting the Presence of Atrial Fibrillation
Acronym: iRead
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: AliveCor (Industry)
Responsible Party: Principal Investigator, Khaldoun Tarakji, Staff, The Cleveland Clinic
Other Study IDs: 14-612
Record Dates: First submitted 2014-08-06; First posted 2014-08-12 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients with Atrial Fibrillation: Patients with Atrial Fibrillation admitted to the hospital for drug loading with Dofetilide or Sotalol willing to record and transmit heart rhythm using AliveCor.
  Interventions: Device: Record and transmit heart rhythm

INTERVENTIONS:
Device: Record and transmit heart rhythm — The patient uses the AliveCor device to record and transmit heart rhythm two times a day. The patient, device software, and Electrophysiologist interpret the rhythm

SUMMARY:
The purpose of this study is to examine whether patients can use the AliveCor case to record their heart rhythm and to assess the accuracy of the software in detecting AF vs sinus rhythm

DETAILED DESCRIPTION:
AliveCor is a new monitoring technology used with a smart phone which allows patients to record their rhythm. The study will compare AliveCor recordings and automated interpretation of the rhythm with the interpretation by an Electrophysiologist.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between > 18 and < 80 years of age
2. Paroxysmal or persistent atrial fibrillation
3. Admitted for antiarrhythmic drug loading (Dofetilide or Sotalol)
4. Already has iPhone 4, 4S or 5 with data plan that accommodates the AliveCor case
5. Willing to use the Alive Cor case
6. Written informed consent

Exclusion Criteria:

1. Unable or unwilling to use the Alive Cor case for their smart phone
2. Presence of a permanent pacemaker

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the hospital for your atrial fibrillation or atrial flutter
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Examine the accuracy of the AliveCor software in detecting AF or sinus rhythm compared to the physician interpretation | 6 month
  Both the software nd overreading electrophysiologist come to the same conclusion regarding the rhythm of the ECG and Alivecor reading. Both determining that the tracing is either normal sinus rhythm or atrial fibrillation.

SECONDARY OUTCOMES:
Assess the correlation between QT interval derived from the AliveCor device compared to standard 12 lead ECG, as assessed by the overreading electrophysiologists. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Khaldoun Tarakji, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] William AD, Kanbour M, Callahan T, Bhargava M, Varma N, Rickard J, Saliba W, Wolski K, Hussein A, Lindsay BD, Wazni OM, Tarakji KG. Assessing the accuracy of an automated atrial fibrillation detection algorithm using smartphone technology: The iREAD Study. Heart Rhythm. 2018 Oct;15(10):1561-1565. doi: 10.1016/j.hrthm.2018.06.037. Epub 2018 Aug 22. PMID 30143448